CLINICAL TRIAL: NCT04949503
Title: A Real-world Study of the Efficacy and Safety of Nimotuzumab in Combination With Chemoradiotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: A Real-world Study of the Efficacy and Safety of Nimotuzumab in Combination With Chemoradiotherapy for LASCCHN
Acronym: Redbull-1
Status: Completed | Type: Observational
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: BPL-Nimo-SCCHN-RWS-1
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — nimotuzumab; Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Patients of study group were all treated with chemoradiotherapy plus nimotuzumab.
  Interventions: Drug: nimotuzumab
- control group: Patients of control group were only treated with chemoradiotherapy, and were collected at least 3 times as many patients as the study group.

INTERVENTIONS:
Drug: nimotuzumab — Patients in the study group were received nimotuzumab on the basis of chemoradiotherapy (control group).
  Other Names: chemoradiotherapy
  Groups: study group

SUMMARY:
This study is a retrospective real-world study. In this study, we plan to collect the clinical data of LASCCHN patients who received chemoradiotherapy combined with or without nimotuzumab .

DETAILED DESCRIPTION:
This study is a retrospective real-world study. The diagnosis and treatment of patients, disease management, and information collection are completely dependent on the daily medical practice. In this study, we plan to select 5 to 8 hospitals nationwide to collect the clinical data of LASCCHN patients who received chemoradiotherapy combined with or without nimotuzumab from January 2015 to December 2018. Patients included in the study will be followed up for survival. The main endpoint is 3-year overall survival (OS) rate; the secondary endpoint are 3-year progression-free survival (PFS) rate, 3-year Local-regional control (LRC) rate, objective response rate (ORR), disease control rate (DCR) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, no gender limitation;
* Histopathologically or cytologically proved to be phase III-IVb of head and neck squamous cell carcinomas (including oral cancer, oropharynx cancer, hypopharynx cancer, larynx cancer, but except for nasopharyngeal carcinoma).
* Patients who received chemoradiotherapy combined with or without nimotuzumab from January 2015 to December 2018;
* Patients in the study group received nimotuzumab, while patients in the control group did not receive nimotuzumab. And patients in the control group were collected 3 times as many cases as the study group in each center. If the number of patients in the control group were less than 3 times of the study group, all cases were collected.

Exclusion Criteria:

* Complicated with primary malignancies other than head and neck tumors (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* Patients received other targeted therapy, immunotherapy, or Traditional Chinese medicine with anti-tumor effect, along with the application of nimotuzumab;
* Lack of critical evaluation information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were more than 18 years old, and were proved to be LASCCHN were included in this study. Patients in the control group receive chemoradiotherapy, while patients in the study group received nimotuzumab on the basis of chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1931 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
3-year overall survival (OS) rate | Up to 3 years
  3-year overall survival (OS) rate

SECONDARY OUTCOMES:
3-year progression-free survival (PFS) rate | Up to 3 years
  3-year progression-free survival (PFS) rate
3-year Local-regional control (LRC) rate | Up to 3 years
  3-year Local-regional control (LRC) rate
objective response rate (ORR) | Up to 12 months
  objective response rate (ORR)=CR+PR
disease control rate (DCR) | Up to 12 months
  disease control rate (DCR)
Safety as measured by number and grade of adverse events | Up to 3 years
  Classification, frequency, and severity of drug-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jinyi Lang, Study Chair — Sichuan Cancer Hospital and Research Institute; Chenping Zhang, Study Chair — Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medcine; Junlin Yi, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Centre, Guangzhou, Guangdong
  - First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shannxi
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality